CLINICAL TRIAL: NCT02420964
Title: Effectiveness of Web-based Teaching to Traditional Patient Education in the Use of Injectable Fertility Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 06-12-10E
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2015-04

CONDITIONS: Infertility
Keywords: injectable; teaching methods
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse instruction (Other): Traditional injection teaching method. No video instruction
  Interventions: Other: Nurse instruction
- Video instruction (Other): Video instruction that can be paused/repeated by subject
  Interventions: Other: video instruction

INTERVENTIONS:
Other: video instruction — Patient Directed Video Instruction
  Arms: Video instruction
Other: Nurse instruction — Nurse directed instruction
  Arms: Nurse instruction

SUMMARY:
The study will be a prospective randomized trial involving human subjects. The study population will consist of all infertility patients presenting to the Carolinas Medical Center Women's Institute who will require injectable use.

Exclusion criteria: Any patient with prior history of IVF injectable use will be excluded from the study.

Independent Variables: The independent variable is the random assignment of each participant to receive either web-based or one on one teaching.

Outcome Variables: The primary outcome variable is the level of knowledge after the intervention. Secondary outcome variables include level of satisfaction with education, preference of educational method, and time required to teach.

Confounding Variables: Potentially confounding variables include age, race, and prior experience with web-based teaching.

DETAILED DESCRIPTION:
Study Design:

The study will be a prospective randomized trial involving human subjects. The study population will consist of all infertility patients presenting to the Carolinas Medical Center Women's Institute who will require injectable use.

Exclusion criteria: Any patient with prior history of IVF injectable use will be excluded from the study.

Independent Variables: The independent variable is the random assignment of each participant to receive either web-based or one on one teaching.

Outcome Variables: The primary outcome variable is the level of knowledge after the intervention. Secondary outcome variables include level of satisfaction with education, preference of educational method, and time required to teach.

Confounding Variables: Potentially confounding variables include age, race, and prior experience with web-based teaching.

Methods:

1. A responsible clinician who has acquainted himself/herself with the research protocol will explain the study to each patient. Patients who agree to participate will sign a form documenting informed consent. The patient will then be handed an envelope that determines whether they will receive web-based teaching or one-on-one teaching.
2. The patients receiving web-based teaching will be taken to a private room to watch a video on injectable medication use. The amount of time required to view the video will be recorded. The video can be paused, rewound and watched as many times as the patient desires.
3. The patients randomized to one-on-one teaching will be taken to a separate room where they will be taught injectable medication use by one of two training healthcare providers with experience teaching injectable medications. The time spent in the teaching session will be recorded.
4. After the teaching session, each patient in the study will complete a multiple choice post-test regarding their knowledge of injectable medication use. They will also complete a satisfaction survey which will use a Likert scale to assess the patients' responses. The instructors teaching the one-on-one sessions will not have access to the post-test.

Statistics:

The categorical variables will be summarized with frequencies and percentages while the continuous variables will be evaluated with means and standard deviations. A difference in proportion will be tested based on the data collected between the web-based group and didactic group. Non-inferiority testing will be conducted based on these differences with a 5% significance level. Data analysis will be conducted using SAS statistical software (9.2,Cary,NC,USA) .

Sample Size Estimate:

To predict that the web-based testing group is not inferior to the Didactic testing group about 40 people in each group would be needed to achieve 80% power with a 5% significance level. The sample size needed was calculated using the Z-test. Here it is assumed that the didactic group would get 80% of their answers correct and the web-based group would actually have 90% of their answers correct.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing ART Therapy and ovulation induction via gonadotropins injection.

Exclusion Criteria:

* Any patient with prior history of IVF injectable use will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Tthe level of knowledge after the intervention measured by a multiple choice post-test | approximately 1 hour
  multiple choice post-test regarding their knowledge of injectable medication use

SECONDARY OUTCOMES:
Satisfaction with education measured by the Likert scale survey | post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center - Women's Institute, Charlotte, North Carolina, United States